CLINICAL TRIAL: NCT02710604
Title: A Phase 2, Randomized, Open-label, Ascending, Sequential Dose Group, Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of CMX157 in HBV-infected Subjects
Brief Title: Phase 2, Multiple Ascending Dose Proof of Concept Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ContraVir Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: ContraVir (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRV-CMX157-201
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2016-12

CONDITIONS: Infectious Disease
Keywords: chronic hepatitis B(CHB)
MeSH Terms: conditions — Communicable Diseases; Hepatitis B, Chronic | interventions — hexadecyloxypropyl 9-(2-(phosphonomethoxy)propyl)adenine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CMX157 5mg versus TDF (Active Comparator): CMX157, 5mg tablet, 28 days versus TDF(tenofovir disoproxil fumerate) 300mg tablet, 28 days
  Interventions: Drug: CMX157; Drug: TDF
- CMX157 10mg versus TDF (Active Comparator): CMX157, 10mg tablet, 28 days versus TDF 300mg tablet, 28 days
  Interventions: Drug: CMX157; Drug: TDF
- CMX157 25mg versus TDF (Active Comparator): CMX157, 25mg tablet, 28 days versus TDF 300mg tablet, 28 days
  Interventions: Drug: CMX157; Drug: TDF
- CMX157 50mg versus TDF (Active Comparator): CMX157, 50mg tablet, 28 days versus TDF 300mg tablet, 28 days
  Interventions: Drug: CMX157; Drug: TDF
- CMX157 100mg versus TDF (Active Comparator): CMX157, 100mg tablet, 28 days versus TDF 300mg tablet, 28 days
  Interventions: Drug: CMX157; Drug: TDF

INTERVENTIONS:
Drug: CMX157 — tablet
  Other Names: lipid conjugate TFV(tenofovir)
Drug: TDF — 300mg tablet
  Other Names: tenofovir disoproxil fumerate

SUMMARY:
This is a phase 2a study to evaluate the safety and tolerability of multiple oral doses of CMX157 at increasing dose levels.

DETAILED DESCRIPTION:
This is a phase 2a study to evaluate the safety and tolerability of multiple oral doses of CMX157 at increasing dose levels in hepatitis B virus(HBV) infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent.
* Capable of completing study requirements.
* Chronic hepatitis B positive.
* HBV treatment naïve.

Exclusion Criteria:

* Positive result for HCV(hepatitis C virus), HDV(hepatitis D virus) or HIV(human immunodeficiency virus).
* History or medical condition that could impact patient safety.
* Current or past abuse of alcohol or illicit drugs.
* Abnormal laboratory value or ECG.
* Pregnant or breastfeeding.
* Clinical, histologic or laboratory evidence of significant liver fibrosis or cirrhosis.
* Systemic immunosuppression.
* Received an investigational drug or investigational vaccine within the 90 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of increasing multiple oral doses of CMX157 in HBV + patients | 28 days
  Capture adverse events, physical examinations, ECGs and clinical laboratory panels
To evaluate the antiviral activity of CMX157 versus tenofovir disproxil fumarate(TDF). | 28 days
  HBV DNA levels

SECONDARY OUTCOMES:
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in HBV + subjects, Cmax. | 28 days
  Measuring Cmax(concentration maximum): the peak plasma concentration.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in HBV + subjects: Tmax. | 28 days
  Measuring Tmax(time maximum): the time Cmax was observed.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in HBV + subjects: AUC. | 28 days
  Measuring AUC(area under the curve): area under plasma concentration versus time curve.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in HBV + subjects: Cmin. | 28 days
  Measuring Cmin(concentration minimum): minimum observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: John Sullivan-Boylai, MD, Study Chair — ContraVir Pharmaceuticals, Inc.
Locations (1):
- Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes